CLINICAL TRIAL: NCT05996770
Title: Evaluation of the Safety and Efficacy of Azvudine and Paxlovid in the Treatment of Hospitalized Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xiao Li，MD (Other)
Responsible Party: Sponsor-Investigator, Xiao Li，MD, Associate professor of pharmacy, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: LCYX-LX-20230102
Record Dates: First submitted 2023-08-16; First posted 2023-08-18 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-11

CONDITIONS: Paxlovid; Azvudine; COVID-19
Keywords: Paxlovid; Azvudine; COVID-19; effectiveness; real-world evidence
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with COVID-19 packaged with Paxlovid: Treatment of patients with COVID-19 with Paxlovid
- Patients with COVID-19 packaged with Azvudine: Treatment of patients with COVID-19 with Azvudine
- Patients with COVID-19 packaged with Paxlovid and Azvudine: Treatment of patients with COVID-19 with Paxlovid and Azvudine

SUMMARY:
In this retrospective study, we aimed to evaluate the clinical efficacy and safety of two antiviral drugs on COVID-19 and inpatients with existing complications in the First Affiliated Hospital of Shandong First Medical University. In addition, we also explored a key issue. Is the combined treatment effect of two antiviral drugs, Paxlovid and Azvudine, better than the use of a single drug?

DETAILED DESCRIPTION:
We conducted a single center retrospective cohort study on hospitalized patients with severe acute respiratory syndrome coronavirus type 2 infection who received treatment with nimatevir/ritonavir tablets or azivudine tablets at the First Affiliated Hospital of Shandong First Medical University from December 1，2022 to January 31，2023. In the research of this project, it is necessary to extract, sort out and retrospectively analyze the clinical data of all patients with COVID-19 who have received Nematovir/Ritonavir tablets or Azivudine tablets in the First Affiliated Hospital of Shandong First Medical University (Shandong Qianfoshan Hospital), and respectively identify the relevant epidemiological characteristics of COVID-19 patients, It is planned to use multiple linear regression or logical regression model to explore the relevant factors that affect the drug use efficiency index, safety index and total cost of patients with COVID-19, so as to provide scientific and quantitative evidence support for the drug use mode of the disease, the clinical value of the drug and the rational drug use of patients, and also provide favorable basis for the supervision and decision-making of smart pharmacy of medical institutions.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient's admission time is from December 1,2022 to January 31,2023. 2. The patient has used either Paxlovid or azivudine tablets during admission. 3. Age ≥ 18 years old. Exclusion Criteria：
* 1. Patients using other antiviral drugs. 2. Patients with incomplete clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All inpatients who were treated with nimatevir/ritonavir tablets and azivudine tablets at the First Affiliated Hospital of Shandong First Medical University from December 1,2022 to January 31,2023.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
mortality | Through study completion，up to half a year.
  Mortality rate of patients with COVID-19 treated with COVID-19 Medicine